CLINICAL TRIAL: NCT05734872
Title: Psychiatry Department of The Second Affiliated Hospital of Zhejiang University School of Medicine
Brief Title: Research on the Intervention of VR-based Emotion Regulation Technology on Adolescent Non-suicide Self-injury Behavior
Acronym: VR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0754
Record Dates: First submitted 2023-02-07; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Non-suicidal Self-injury
Keywords: Non-suicidal Self-injury; Virtual Reality Technology; Adolescent
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Device: Virtual Reality Technology
- Control group (Other)
  Interventions: Other: Routine mental health course training

INTERVENTIONS:
Device: Virtual Reality Technology — Make a pair of glasses through virtual reality technology, through which participants can observe and participate in the treatment process.
  Arms: Experimental group
Other: Routine mental health course training — Conduct mental health education for patients by making a speech.
  Arms: Control group

SUMMARY:
Non suicidal self injury (NSSI) has become a serious social and public health problem allover the world, and the incidence rate is increasing year by year. Although the aim of NSSI is not to suicide, but its negative impact is extremely serious, which will seriously threaten the physical and mental health of adolescents. Virtual Reality (VR), a computer simulation technology, can enable people to enter and experience the artificial virtual world in an immersive way, has been used for the auxiliary treatment of anxiety disorder, post-traumatic stress disorder and other diseases. This study explored the impact of VR on the depression and mental health of NSSI adolescents, so as to reduce the incidence of non-suicide self-injury behavior in NSSI adolescent patients and improve the quality of life of such patients.

ELIGIBILITY:
Inclusion Criteria:

* According to the diagnostic criteria of NSSI in the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders.
* Have a past history of non-suicidal self-injury behavior.
* No virtual reality technology intervention before enrollment.
* age: ≥ 18 to<24.

Exclusion Criteria:

* Those who have serious physical diseases
* Those who cannot cooperate with the completion of virtual reality technology finally complete the intervention content<50%.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-12-26 (Estimated); Study Completion 2024-10-26 (Estimated)

PRIMARY OUTCOMES:
Ottawa Self-injury Inventory Chinese Revision | up to one month
  This item describes the addictive characteristics of non-suicidal self-injury behavior. There are seven items in total. Add the seven items to get the original total score. The higher the original total score, the more addictive the non-suicidal self-injury behavior of the individual. The minimum value is 0 and maximum value is 28.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Chen, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China